CLINICAL TRIAL: NCT04150640
Title: Phase 2 Trial of 5-Fluorouracil, Oxaliplatin and Liposomal Irinotecan and Immunotherapy (Plus Trastuzumab for HER2-positive Disease) During 1st Line Treatment of Advanced Esophageal and Gastric Adenocarcinoma
Brief Title: Oxaliplatin and Liposomal Irinotecan (Plus Trastuzumab for HER2-positive Disease) in Advanced Esophageal and Gastric Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW19029; NCI-2019-07966 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); 2019-0632 (Other: Institutional Review Board); Protocol Version 7/1/2024 (Other: UW Madison)
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Adenocarcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Trastuzumab; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: HER2 Negative (Experimental): Participants in Cohort 1 (HER2-negative) will be treated with nal-IRI (50 mg/m^2 - intravenously over 90 min), 5-FU (2400 mg/m^2 over 46 hrs), and oxaliplatin (60 mg/m^2). Each cycle is 28 days. Participants will receive treatments on day 1 and 15 of each cycle.
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: 5-FU
- Cohort 2: HER2 Positive (Experimental): Participants in Cohort 2 (HER2-positive) will be treated with nal-IRI (50 mg/m^2 - intravenously over 90 min), trastuzumab (6 mg/kg C1D1, then 4 mg/kg on each subsequent treatment days), 5-FU (2400 mg/m^2 over 46 hrs), and oxaliplatin (60 mg/m^2). Each cycle is 28 days. Participants will receive treatments on day 1 and 15 of each cycle.
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: 5-FU; Drug: Trastuzumab
- Cohort 3: HER2 Negative (Experimental): Participants in Cohort 3 (HER2-negative) will be treated with nal-IRI (50 mg/m^2 - intravenously over 90 min), 5-FU (2400 mg/m^2 over 46 hrs), oxaliplatin (60 mg/m^2), and nivolumab. (240 mg). Each cycle is 28 days. Participants will receive treatments on day 1 and 15 of each cycle
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: 5-FU; Drug: Nivolumab
- Cohort 4: HER2 Positive (Experimental): Participants in Cohort 4 (HER2-positive) will be treated with nal-IRI (50 mg/m^2 - intravenously over 90 min), trastuzumab (6 mg/kg C1D1, then 4 mg/kg on each subsequent treatment days), 5-FU (2400 mg/m^2 over 46 hrs), oxaliplatin (60 mg/m^2), and pembrolizumab (400 mg). Each cycle is 42 days. Participants will receive chemotherapy and trastuzumab treatments on day 1, 15, and 29 of each cycle. Pembrolizumab will be given on day 1 of each cycle.
  Interventions: Drug: Nal-IRI; Drug: Oxaliplatin; Drug: 5-FU; Drug: Trastuzumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nal-IRI — chemotherapy drug
  Other Names: liposomal irinotecan
Drug: Oxaliplatin — chemotherapy drug
Drug: 5-FU — chemotherapy drug
  Other Names: Fluorouracil
Drug: Trastuzumab — immunotherapy
  Arms: Cohort 2: HER2 Positive; Cohort 4: HER2 Positive
Drug: Pembrolizumab — immunotherapy
  Arms: Cohort 4: HER2 Positive
Drug: Nivolumab — immunotherapy
  Arms: Cohort 3: HER2 Negative

SUMMARY:
This is an open label, phase II, multi-site trial evaluating the efficacy and safety of the combination of 5-FU, oxaliplatin, nal-IRI, and immunotherapy (plus trastuzumab for HER2-positive tumors) as first-line therapy for participants with advanced Esophageal and Gastric Adenocarcinoma (EGA). The investigators hypothesize that this drug combination will be better tolerated than current first-line chemotherapy combinations for this disease.

DETAILED DESCRIPTION:
This is an open label, phase II, multi-site trial evaluating the efficacy and safety of the combination of 5-FU, oxaliplatin, nal-IRI, and immunotherapy (plus trastuzumab for HER2-positive tumors) as first-line therapy for participants with advanced Esophageal and Gastric Adenocarcinoma (EGA).

Participants will be enrolled into one of four cohorts. Participants in Cohort 1 (HER-2 negative) will receive 5-FU, oxaliplatin and nal-IRI. Cohort 3 (HER-2 negative) will use nivolumab in addition to 5-FU, oxaliplatin and nal-IRI. Participants in Cohort 2 (HER-2 positive) will receive trastuzumab in addition to 5-FU, oxaliplatin and nal-IRI. Cohort 4 (HER-2 positive) will also include pembrolizumab in addition to trastuzumab, 5-FU, oxaliplatin and nal-IRI.

Chemotherapy doses will be the same for all cohorts and will follow similar modifications for toxicities. Agents will be administered as per institutional standards when similar regimens (such as FOLFIRINOX, FOLFOX, and trastuzumab) are used.

Cohort 1 (HER2-negative tumors): Up to 13 evaluable participants will be accrued to Cohort 1.

Cohort 2 (HER2-positive tumors): Up to a total of 6 subjects will be enrolled to evaluate the safety and tolerability of the proposed 5-Fluorouracil, Oxaliplatin and liposomal Irinotecan combination in HER2-positive subjects.

Cohort 3 (HER-2 negative tumors):12 participants will be enrolled during stage 1. If at most 5 objective responses per RECIST 1.1 are observed, then further enrollment will be halted. Otherwise, 15 additional participants will be enrolled for a total number of 27.

Cohort 4 (HER-2 positive tumors): treated with oxaliplatin, Nal-IRI and trastuzumab in combination with pembrolizumab. A total of up to 6 subjects will be accrued to evaluate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.

NOTE: HIPAA authorization may be included in the informed consent or obtained separately.

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Histological or cytological confirmed locally advanced or metastatic EGA. Known HER2 status prior to treatment initiation required. Known PDL1 CPS status prior to treatment initiation.
* Measurable disease according to RECIST v1.1.
* No prior lines of systemic therapy for advanced disease.
* Participants who had received neoadjuvant or adjuvant therapy or definitive chemoradiation will be allowed to participate if recurrence occurred 6 months or longer from the completion of all prior treatments.
* Demonstrate adequate organ function as defined below; all screening labs to be obtained within 14 days prior to registration

  * Absolute Neutrophil Count (ANC) ≥1,500 /μl without the use of hematopoietic growth factors
  * Hemoglobin (Hgb) ≥8 g/dL (blood transfusions are permitted for participants with hemoglobin levels below 8 g/dL)
  * Platelets ≥100,000 /μl
  * Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl). CrCl calculation using the Cockcroft-Gault formula. ≥50 mL/min for participants with creatinine levels > 1.5 X institutional ULN
  * Bilirubin within normal range for the institution (biliary drainage is allowed for biliary obstruction)
  * Aspartate aminotransferase (AST) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Alanine aminotransferase (ALT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >3.0 g/dL
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Women of childbearing potential should have a negative urine or serum pregnancy test within 14 days of study registration. NOTE: Women are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Women of childbearing potential and males must be willing to abstain from heterosexual activity or to use a form of effective method of contraception from the time of informed consent until 30 days after treatment discontinuation.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Known hypersensitivity to 5-FU, oxaliplatin or other platinum agents, or any of the components of nal-IRI and other liposomal products.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency (testing not required prior to enrollment).
* Other active malignancy requiring treatment within the last 2 years. Exceptions include subjects with non-melanoma skin cancer, non-invasive/in situ cancer or low-risk prostate cancer requiring hormonal therapy only.
* Current therapy with other investigational agents or participation in another clinical study (supportive care and nontherapeutic trial participation allowed if not receiving an investigational drug). Participants may participate in prescreening for other therapeutic trials (prescreening of biologic sample for specific mutations, receptors, etc.)
* Major surgery within 28 days or minor surgery within 14 days of the start of the study treatment, except for tumor biopsy or placement of central infusion device (port placement).
* Radiotherapy less than 7 days prior to the start of the study treatment
* Participants who receive nivolumab or pembrolizumab in addition to chemotherapy should not have any contraindications to immune checkpoint inhibitors and should not have received immunotherapy agents for the treatment of EGA prior to study enrollment.

  * Participants must not have active autoimmune disease that has required systemic treatment in the past 2 years. Participants are permitted to receive immunotherapy l if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
  * Participants must not have a condition requiring systemic treatment with either corticosteroids (>10 mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of study immunotherapy administration. Inhaled or topical steroids and adrenal replacement doses (≤10 mg/day prednisone equivalent) are permitted. Participants with prior immune mediated adverse events related to immunotherapy that resulted in permanent treatment discontinuation with these agents.
* Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.
* Active infection requiring systemic therapy.
* Pregnant or breastfeeding.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before inclusion.
* NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure.
* Known history of Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Objective Response Rate (ORR) | up to 1 year
  ORR will be calculated by combining the number of participants who achieve complete response and partial response per RECIST 1.1 criteria, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment). An ORR of 40% or less for proposed combination of 5-Fluorouracil, Oxaliplatin and nal-IRI during 1st line treatment of advanced esophageal and gastric adenocarcinoma in HER2-negative subjects will be considered as unacceptably low. The number and frequencies of objectives responses will be summarized in tabular format. The ORR will be reported along with the corresponding one-sided 90% confidence intervals.
Cohort 3: Objective Response Rate (ORR) | up to 1 year
  ORR will be calculated by combining the number of participants who achieve complete response and partial response per RECIST 1.1 criteria, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment). An ORR of 45% or less for proposed combination of 5-Fluorouracil, Oxaliplatin, nal-IRI and Nivolumab during 1st line treatment of advanced esophageal and gastric adenocarcinoma in HER2-negative subjects will be considered as unacceptably low. The number and frequencies of objectives responses will be summarized in tabular format. The ORR will be reported along with the corresponding one-sided 90% confidence intervals.
Cohorts 2 and 4: Incidence of Adverse Events | up to 1 year
  The primary objective of cohorts 2 and 4 (HER2-positive EGA) is to evaluate safety and tolerability of the studied drug combination. Toxicities and adverse events will be summarized by type and severity in tabular format.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 2 years
  PFS will be defined from the date study enrollment to the date of progression event or death. If a participant does not experience a progression event at the end of the follow-up period, then the PFS will be censored at the last assessment date. PFS will be analyzed using the Kaplan-Meier method. Median PFS will be reported along with the corresponding 90% confidence interval which will be constructed using the nonparametric Brookmeyer-Crooley method.
Disease Control Rate (DCR) | up to 1 year
  The DCR is the proportion of all participants with stable disease (SD) for 8 weeks, or partial response (PR), or complete response (CR) according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).DCR will be reported along with the corresponding 90% confidence intervals which will be constructed using the Wilson score method.
Progression Free Survival at 6 months | up to 6 months
  PFS will be defined from the date study enrollment to the date of progression event or death. If a participant does not experience a progression event at the end of the follow-up period, then the PFS will be censored at the last assessment date. PFS will be analyzed using the Kaplan-Meier method. Median PFS will be reported along with the corresponding 90% confidence interval which will be constructed using the nonparametric Brookmeyer-Crooley method.
Progression Free Survival at 12 months | up to 1 year
  PFS will be defined from the date study enrollment to the date of progression event or death. If a participant does not experience a progression event at the end of the follow-up period, then the PFS will be censored at the last assessment date. PFS will be analyzed using the Kaplan-Meier method. Median PFS will be reported along with the corresponding 90% confidence interval which will be constructed using the nonparametric Brookmeyer-Crooley method.
Cohorts 1 and 3: Incidence of Adverse Events | up to 1 year
  Toxicities and adverse events will be summarized in tabular format, stratified by type and severity
Cohorts 2 and 4: Overall Response Rate | up to 1 year
  ORR will be calculated by combining the number of participants who achieve complete response and partial response per RECIST 1.1 criteria, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Uboha, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu